CLINICAL TRIAL: NCT02367807
Title: Pre-Exposure Prophylaxis With TDF/FTC to Prevent HIV-1 Acquisition in Young Men and Transgender Women of Color Who Have Sex With Men
Brief Title: PrEP With TDF/FTC to Prevent HIV-1 Acquisition in Young MSM and Transgender Women of Color
Status: Completed | Type: Observational
Sponsor: Philadelphia Fight (Other)
Responsible Party: Sponsor
Other Study IDs: IN-US-276-1295
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: HIV
Keywords: HIV prevention; PrEP; young men who have sex with men; Truvada
MeSH Terms: interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine and plasma samples for measurement of tenofovir concentration, blood samples for measurement of safety labs, and urine/plasma samples and rectal/pharyngeal swabs for sexually transmitted infection screening
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Emtricitabine and tenofovir disoproxil fumarate — This study will enroll 50 subjects who are offered TDF/FTC for 48 weeks as part of a combined biomedical/behavioral intervention offered in a community-based setting serving high-risk youth in an urban setting.
  Other Names: Truvada; TDF/FTC

SUMMARY:
This is a 48-week prospective observational study that will allow testing of the hypothesis that a program in which pre-exposure prophylaxis (PrEP) is administered to young men of color who have sex with men (yMSMc) in a community youth drop-in center in conjunction with a multifaceted behavioral intervention as well as standard HIV prevention interventions can achieve at least 70% retention, as well as a medication adherence rate significantly better than that previously reported in the literature. The proposed program evaluation can provide critical information for the enhancement and scale-up of successful PrEP programs at FIGHT and elsewhere in an effort to make PrEP available to a growing number of persons at risk of acquiring human immunodeficiency virus (HIV).

DETAILED DESCRIPTION:
PrEP for HIV prevention with once daily Truvada has been shown to be extremely safe and efficacious in multiple populations when taken consistently. Young men who have sex with men of color (yMSMc) comprise the group at the highest risk of new HIV infections and the only group whose HIV infection rates continue to increase. New data suggest interrupting transmission among MSM can reduce HIV acquisition among other risk groups as well. However, accessing, linking, and retaining yMSMc in a PrEP program is both critical to successful HIV prevention and historically difficult to achieve. Philadelphia FIGHT initiated a PrEP program at the youth site, Youth Health Empowerment Project (Y-HEP), for yMSMc approximately 1.5 years ago that also gives all participants access to general primary care. Y-HEP utilizes a unique biomedical/biobehavioral approach to enhance adherence and retention of yMSMc receiving PrEP.

The purpose of this protocol is to increase access to safe and effective PrEP to yMSMc in order to reduce incident HIV infections and health disparities in HIV incidence and prevalence through the use of a combined biomedical/behavioral intervention in a community-based setting servicing high-risk youth in Philadelphia. It is hypothesized this unique, combined biomedical/behavioral HIV prevention strategy will lead to high recruitment and retention rates in this community setting. All subjects will be offered primary care services as well as a package of HIV risk reduction interventions including once daily PrEP with tenofovir and emtricitabine (TDF/FTC), condoms, risk reduction counseling, HIV testing, and sexually transmitted infection (STI) screening and treatment. A weekly support group will aim to maximize medication adherence and retention by engaging subjects in prevention, risk-reduction and behavioral counseling, education about HIV, leadership training, and social networking.

Subjects will consist of 50 HIV-negative biological males between the ages of 18 and 30 who meet eligibility criteria as defined below.

All subjects will receive Truvada as PrEP on Monday evenings on an either weekly, biweekly, or monthly basis depending on an initial assessment of their need for adherence support, with provisions to obtain medication the following day(s) at Y-HEP if they are unable to attend the Monday night session. Study subjects will be considered to have picked up their medications if they come any time during the week designated as a medication pick-up week. In addition, all subjects will receive standard HIV prevention services including condom provision, risk reduction counseling, HIV testing, STI screening and treatment, as well as basic medical care and linkage to HIV care in the event of PrEP failure. Subjects will receive a behavioral intervention consisting of youth-focused men's wellness services centered around education about HIV, adherence counseling and knowledge of PrEP efficacy on risk behavior, general health services such as smoking cessation support and nutritional counseling, job and leadership training, and sexual health and well-being promotion.

Subjects will be screened for HIV, STIs, and renal function at baseline and every three months, and will also have a rapid test for HIV on a monthly basis (Table 1). Treatment will be provided for all STIs diagnosed during this study, and non-immune subjects will be offered vaccines against hepatitis A and B. Adherence will be assessed by the percentage of medication pick-up visits attended as well as urine tenofovir levels every 2-4 weeks and plasma tenofovir levels at weeks 24 and 48. Risk behaviors will be assessed by STI rates and the adapted Risk Assessment Battery at baseline, and weeks 24 and 48. A qualitative interview will be conducted at the end of the study to assess program acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 30 years at the time of signed informed consent
* Willing and able to independently provide written informed consent
* Biological male at birth
* Tests HIV negative at time of screening using rapid HIV antibody test (HIV viral load testing is also conducted immediately prior to initiation of PrEP, but is not an inclusion criteria as screening labs may be collected weeks prior to medication initiation and we would like to confirm a negative viral load as close to medication initiation as possible for subject's safety)
* Willing to provide locator information to study staff for a 48-week period
* Current participant in I Am Men's Health PrEP program or willing to become a participant

Exclusion Criteria:

* Evidence of acute or chronic hepatitis B infection at the time of screening
* Other clinically significant acute or chronic medical condition, including severe infections requiring treatment such as tuberculosis, as determined by the study investigator
* Evidence of renal dysfunction (Creatinine Clearance < 50 ml/min) at the time of screening; Use Cockcroft-Gault equation: GFR = (140-Age in years) x (Weight in kg) / (72 x serum creatinine)
* History of bone fractures not explained by trauma
* Grade 3 laboratory abnormality on screening tests/assessments as defined by the DAIDS grading system
* Concurrent participation in an HIV vaccine study
* Known allergy/sensitivity to the study drug or its components
* Current use of any antiretroviral agent other than Truvada for any reason
* Experiencing decompensated cirrhosis (e.g., ascites, encephalopathy, etc.)
* Any other clinical condition or prior therapy that, in the opinion of the Principal Investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50 biological males from urban Philadelphia who identify as men who have sex with men (MSM) ages 18-30 at risk of HIV acquisition
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Evaluate program retention | 48 weeks
  We will determine whether this community intervention can achieve 70% program retention at the end of 48 weeks, as defined by the proportion of patients initiating Truvada who pick up at least 50% of their medication through 48 weeks and who have a study visit in the 48-week window (subject may have this final study visit within an allowed window of 4 weeks before or after the 48-week visit in accordance with the FDA snapshot algorithm). Intermediate retention assessment will also be conducted at weeks 12, 24, and 36 by assessing the proportion of patients who have picked up at least 50% of their medication prior to those time points and who have a study visit at the end of those periods using +/- 4 week snapshot analysis.
Evaluate adherence to PrEP | 48 weeks
  This will be assessed by the proportion of medication pick-up visits attended (a function of pharmacy refill data), and the proportion of study subjects with detectable urine drug concentrations over the 48 week study period. We will compare the estimates of adherence obtained with these measurements to two plasma tenofovir concentrations (collected at weeks 24 and 48) using the cutoff of 16 fmol/106 cells as the level associated with 90% adherence or greater.

SECONDARY OUTCOMES:
Assess behavioral change | 48 weeks
  This will be assessed through the change in reported number of risk behaviors at weeks 0, 24 and 48 (as measured by the Risk Assessment Battery, RAB) as well as the change in incidence of STIs over the study period. The RAB provides a brief self-report measure of drug use practices and sexual behaviors associated with HIV transmission. The RAB was developed and validated by the University of Pennsylvania and has been adapted for use in many countries. Study-specific questions in addition to the RAB will focus on attitudes regarding the effect of PrEP on risk behaviors.
Measure program acceptability and feasibility | 48 weeks
  Program acceptability and feasibility will be measured objectively by assessing program retention as well as subjectively through qualitative assessment. A standard acceptability survey adapted from the "HIV Treatment Satisfaction Questionnaire" © Prof. Clare Bradley: 7/97 English for UK & USA rev.12.2.01A (intro.rev.1.10.04), Health Psychology Research, Dept of Psychology, Royal Holloway, University of London, Egham, Surrey, TW20 0EX. UK will be administered to study subjects at the end of the trial (included as attachment of full protocol).
Measure the success rate in linking to care participants who seroconvert to HIV positive status while receiving PrEP | 48 weeks
  This will be measured by the proportion of subjects who seroconvert to HIV positive status during the 48-week study who are seen by an HIV clinician within one week of diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Koenig, MD, MPH, Principal Investigator — Philadelphia Fight
Locations (1):
- Philadelphia FIGHT, Philadelphia, Pennsylvania, United States